CLINICAL TRIAL: NCT04677153
Title: Rapid HCV Test and Treat to Increase HCV Treatment Uptake Among People Who Use Drugs
Brief Title: Rapid HCV Treatment Access for Persons Who Use Drugs
Acronym: RAPID-HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00265240
Record Dates: First submitted 2020-12-17; First posted 2020-12-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hepatitis C Virus Infection, Response to Therapy of
MeSH Terms: conditions — Hepatitis C | interventions — Coal Tar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test and Treat plus Peer Mentors Intervention Arm (Experimental): Participants offered 8 weeks of glecaprevir/pibrentasvir (GLE/PIB) at OTP plus peer support.
  Interventions: Other: Test and treat plus peer mentors
- Standard of Care Referral Arm (Active Comparator): Participants referred to offsite (non-OTP) location for HCV treatment.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Test and treat plus peer mentors — Rapid start of HCV treatment at OTP within days of HCV diagnosis. Participants will receive 8 weeks of glecaprevir/pibrentasvir and will work with a peer mentor during and after treatment.
  Other Names: On-site treatment with peer support HCV treatment implementation strategy
  Arms: Test and Treat plus Peer Mentors Intervention Arm
Other: Usual care — Participants are referred to another location for HCV treatment.
  Other Names: Standard of care referral HCV treatment implementation strategy
  Arms: Standard of Care Referral Arm

SUMMARY:
This study is being done to compare two strategies to deliver HCV treatment to persons with hepatitis C virus (HCV) who also use drugs and are participating in an outpatient opioid treatment program (OTP). Participants will be randomized into one of two treatment groups:

1. Test and treat plus peer-mentors: This treatment group will be offered 8 weeks of glecaprevir/pibrentasvir (an FDA approved HCV treatment) within days of HCV diagnosis at the OTP. Participants in this group will receive treatment adherence support from a peer-mentor who is someone who has been cured of HCV infection.
2. Standard of care HCV treatment referral: This treatment group will be referred to an offsite HCV treatment location. This is the usual care for anyone who tests positive for HCV at the OTP who is not participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness of participant to provide written informed consent
* Men and women age ≥18 to ≤70 years at study entry
* HCV antibody positive/detectable HCV RNA
* HCV treatment naïve (no prior treatment with an approved or investigational oral Direct-Acting Antivirals (DAA) therapy
* Negative pregnancy test at screening or at the day of treatment initiation (females of childbearing potential only)
* If co-infection with Human Immunodeficiency Virus (HIV) is documented, the subject must be anti-retroviral treatment (ART) naïve with CD4 T cell count >500 cells/mm3 OR on a stable ART regimen (containing only permissible ART - Raltegravir; dolutegravir; Rilpivirine; Elvitegravir/cobicistat; Tenofovir disoproxil fumarate; Tenofovir alafenamide; Emtricitabine; Lamivudine and/or Abacavir, bictegravir)

Exclusion Criteria:

* Women who are pregnant or breastfeeding, or considering becoming pregnant during the study and for 30 days after the last dose of study drug
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation
* Current or history of decompensated liver disease (including but not limited to encephalopathy, variceal bleeding, or ascites) prior to study entry
* History of hepatocellular carcinoma (HCC)
* Any history of active Hepatitis B or positive HBsAg test
* Platelet count < 150,000/mm3
* HCV RNA undetectable
* History of clinically significant abnormalities or co-morbidities that make the subject an unsuitable candidate for this study, in the opinion of the investigator.
* Women of childbearing potential that are not practicing at least one specified method of birth control that is effective from Study Day 1 through at least 30 days after the last dose of study drug.
* Subject is currently taking any of the following prohibited medications: red yeast rice (monacolin K), St. John's Wort, carbamazepine, dabigatran, efavirenz, phenytoin, pentobarbital, phenobarbital, primidone, rifabutin, rifampin.
* Subject is not able or willing to safely discontinue the prohibited medications or supplements listed below at least 14 days prior to the first dose of GLE/PIB: some HMG-CoA reductase inhibitors, astemizole, cisapride, terfenadine, ethinyl estradiol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Participants Who Initiate HCV Therapy | Within 12 weeks of randomization
  Proportion of participants who start HCV treatment in each arm.

SECONDARY OUTCOMES:
HCV Treatment Completion | At expected end of treatment date, up to 20 weeks
  Proportion of participants who start HCV treatment and subsequently complete treatment (take more than 90% of prescribed treatment course).
Sustained Virologic Response (SVR) Following Treatment by Intervention Group | Post-treatment week 12
  Proportion of participants in each arm who achieved SVR, defined as HCV RNA <15 IU/mL between 10 and 36 weeks weeks after completion of the HCV treatment regimen.
Time to HCV Treatment Initiation | From randomization to initiation of treatment, up to 24 weeks
  Time to HCV Treatment Initiation in weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwaseun Falade-Nwulia, MBBS, MPH, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
- University Health Network Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No